CLINICAL TRIAL: NCT05138705
Title: An Open Phase IV Clinical Trial of Quadrivalent Influenza Virus Split Vaccine to Evaluate the Safety and Immunogenicity in Healthy Population Aged 3-8 Years
Brief Title: Clinical Trial of Quadrivalent Influenza Virus Split Vaccine in Population Aged 3-8 Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021S00207-01
Record Dates: First submitted 2021-11-28; First posted 2021-12-01 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2021-11

CONDITIONS: Influenza, Human
Keywords: QIV, safety, immunogenicity
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Subjects in one group received a first and a second dose of the vaccine at different time points.
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Outcome (Experimental): Quadrivalent influenza vaccine Participants randomized to receive two injections of 0.5 mL quadrivalent influenza vaccine at Day 0 and 28.
  Interventions: Biological: Quadrivalent Influenza Virus Split Vaccine

INTERVENTIONS:
Biological: Quadrivalent Influenza Virus Split Vaccine — 0.5ml Quadrivalent influenza vaccine The inactivated split virion vaccines contained 15 μg of each hemagglutinin antigen of influenza A/H1N1, A/ H3N2, B/Victoria and B/Yamagata strains

SUMMARY:
To evaluate the safety and immunogenicity of quadrivalent influenza virus split vaccine in healthy population aged 3-8 years following different immunization procedures.

DETAILED DESCRIPTION:
To evaluate the safety and immunogenicity of quadrivalent influenza virus split vaccine in healthy population aged 3-8 years following different immunization procedures, and the participants randomized to receive two injections of 0.5 mL quadrivalent influenza vaccine at day 0 and 28.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 3-8 years. Volunteers are required to show vaccination certificate if they have not received a previous flu vaccine.
* Volunteers' legal guardian or client informed consent, voluntarily participate in and sign informed consent. (Volunteers over the age of 8 also need informed consent and signature)
* Volunteers' legal guardian or client has the ability (non-illiterate) to understand the study procedures, to use a thermometer, scale, and fill in a diary card as required, and be able to complete the clinical study in compliance with the clinical trial protocol.

Exclusion Criteria:

* The axillary temperature greater than 37.0℃ on the day of enrollment;
* Have suffered from influenza within previous 3 months or suffering currently (confirmed by either clinical, serological or microbiological methods);
* Have received any influenza vaccine (registered or experimental) within 6 months or be going to receive other influenza vaccine during the study period;
* Allergic to any component of the vaccine, or have a history of allergic reactions to gentamicin sulfate;
* A history of severe allergy to any vaccine or drug, or with a history of nervous system damage;
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc;
* Acute illness, severe chronic illness or acute attack of chronic disease on the day of vaccination;
* A history of live attenuated vaccination within 14 days prior to vaccination and a history of other vaccinations within 7 days prior to vaccination;
* Received immunoenhancement or inhibitor therapy within 3 months (continued oral or intravenous administration for more than 14 days);
* Congenital or acquired immune deficiency, HIV infection, lymphoma, leukemia or other autoimmune diseases;
* Have a history of asthma, the condition has been unstable for past two years and require treatment, such as emergency treatment, hospitalization, intubation or oral or intravenous administration of corticosteroids and so on;
* Have received blood or blood-related products;
* A history of convulsion, epilepsy, encephalopathy, guillain-barre syndrome, a history of mental illness or have a mental illness family history;
* A history of abnormal coagulation function (such as coagulation factor deficiency, coagulation disease);
* Planning to relocate before the end of the study or to leave for an extended period during the scheduled study visit;
* Participating in or planning to participate in other clinical trials in the near future;
* Any conditions judged by investigators that were inappropriate for participation in this clinical trial.

Receiving the second dose of vaccine

* Have a severe allergic reaction after receiving the first dose of vaccine;
* Serious adverse events occurred that were causally related to the first dose of vaccine injection；
* After receiving the first dose of vaccine, the researchers will decide whether the volunteer should participate in the study continued or not if the newly discovered feature or newly condition occurred on volunteer that do not meet the inclusion criteria or meet the exclusion criteria;
* Other reasons for exclusion considered by the investigator.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 380 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
seroconversion rate of hemagglutination inhibition (HI) antibodies | up to 56 days
  28 days after receiving one and two doses of vaccine in subjects aged 3-8 years, respectively. Seroconversion rate of HI antibodies against any subtype of influenza virus in each group.
seroprotection rate of HI antibodies | up to 56 days
  28 days after receiving one and two doses of vaccine in subjects aged 3-8 years, respectively. Seroprotection rate of HI antibodies against any subtype of influenza virus in each group.
geometric mean increase (GMI) of HI antibodies | up to 56 days
  28 days after receiving one and two doses of vaccine in subjects aged 3-8 years, respectively. GMI of HI antibodies against any subtype of influenza virus in each group.
The proportion of all adverse reactions/events | up to 56 days
  The proportion of all adverse reactions/events in subjects through 28 days after the second dose.

SECONDARY OUTCOMES:
p value of difference of seroconversion rate in subjects with different immunization procedures | up to 56 days
  p value of the difference of seroconversion rate of HI antibodies at 28 days between subjects receiving one dose of vaccine and subjects receiving two.
p value of difference of seroprotection rate in subjects with different immunization procedures | up to 56 days
  p value of the difference of seroprotection rate of HI antibodies at 28 days between subjects receiving one dose of vaccine and subjects receiving two.
p value of difference of GMI in subjects with different immunization procedures | up to 56 days
  p value of the difference of GMI of HI antibodies at 28 days between subjects receiving one dose of vaccine and subjects receiving two.
Reactogenicity Events | 208 days
  The proportion of all adverse reactions/events in subjects from the day subjects receiving the first dose of vaccine to 180 days after subjects receiving the second dose.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Principal Investigator — Shandong Provincial Center for Disease Control and Prevention
Locations (1):
- Tingting and Yu, Tai’an, Shandong, China

IPD SHARING:
Plan to Share IPD: No